CLINICAL TRIAL: NCT00410540
Title: A Randomized, Double-Blind, Controlled Trial of Hydromorphone (Immediate and Sustained- Release) vs Morphine (Immediate and Sustained-release) in Cancer Pain
Brief Title: A Study of OROS Hydromorphone HCL vs Morphine in Cancer Pain Patients.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alza Corporation, DE, USA (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR013261
Record Dates: First submitted 2006-12-12; First posted 2006-12-13 (Estimated); Last update posted 2010-04-27 (Estimated); Status verified 2010-04

CONDITIONS: Pain; Analgesics, Opioid
Keywords: Cancer pain; Oral analgesic; OROS hydromorphone HCL; Morphine sulfate
MeSH Terms: conditions — Pain; Cancer Pain | interventions — Morphine

INTERVENTIONS:
Drug: OROS hydromorphone HCL ; Morphine sulfate

SUMMARY:
The purpose of this study was to demonstrate the clinical equivalence of hydromorphone and morphine (immediate-release [IR] and sustained-release [SR] formulations) using the "worst pain in the past 24 hours" item of the Brief Pain Inventory (BPI). The secondary objective of this study was to compare hydromorphone and morphine in the following variables: other pain measures, various questionnaires, and safety and tolerability variables.

DETAILED DESCRIPTION:
This was a phase-3, multicenter, multinational, randomized (patients are assigned different treatments based on chance), active-controlled, double-blind, multiple-ascending-dose, parallel-group study in adult patients with cancer pain who receive and/or require strong oral or transdermal opioid analgesics (60-540 mg of oral morphine equivalents daily). This study consisted of 2 phases: an initial immediate release (IR) phase and a subsequent slow release (SR) phase. Eligible patients were randomized 1:1 to receive either OROS hydromorphone HCl or morphine sulfate (immediate release formulation in the immediate release phase, slow release formulation in the slow release phase). In the immediate release phase (2-9 days), patients were started on the appropriate initial dose of immediate release medication every 4 hours (q4h), (6 doses/day) using a 5:1 conversion ratio (morphine equivalents:hydromorphone dosage). If the patient had greater than 3 breakthrough-pain episodes requiring additional pain medication in 24 hours, the study medication dosage was increased, at most once a day. When the patient had achieved dose-stable pain control (2 days with 3 or less than 3 breakthrough-pain episodes per day), the patient was permitted to continue into the slow release phase. The patient was given an equivalent dosage of a slow release formulation of the same drug (OROS® hydromorphone HCL each day or morphine sulfate slow release two times per day), administered using a double-dummy technique. Dosage increases were permitted every 2 days if the patient had more than 3 breakthrough-pain episodes in 24 hours. To complete the slow release phase, patients had to achieve dose-stable pain control for at least 2 days.Safety assessments of physical examination, labs and adverse event reporting were done. OROS hydromorphone HCL slow release 8, 16, 32, and 64mg tablets; Morphine sulfate immediate release10, 20, 50 mg capsules;Morphine sulfate slow release 5, 30, 60, 90, 120, 160, and 200mg capsules;hydromorphone immediate release 2, 4, 8 mg;The immediate release medications orally every 4 hours;The OROS hydromorphone slow release formulation orally every 24 hours and morphine slow release orally twice daily.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cancer pain who are currently receiving strong oral or transdermal opioid analgesics or in whom strong opioid analgesics are appropriate
* Patients who requires or are expected to require between 60 and 540 mg of oral morphine or morphine equivalents every 24 hours for the chronic management of cancer pain
* Patients who have pain suitable for treatment with a once-daily formulation
* Patients with concomitant chemotherapy or radiotherapy. Exclusion Criteria:
* Patient with gastrointestinal (GI) disease of sufficient severity to interfere with orally administered analgesia (eg dysphagia, vomiting, constipation, bowel obstruction, severe gut narrowing) were not permitted to enroll
* Patient where the risks of treatment with morphine or hydromorphone outweighed the potential benefits such as raised intracranial pressure, hypotension, hypothyroidism, asthma, reduced respiratory reserve, prostatic hypertrophy, hepatic or renal impairment, convulsive disorders, and Addison's disease
* Debilitated patients were excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Study Completion 2001-05 (Actual)

PRIMARY OUTCOMES:
The primary efficacy : Patient's assessment of "worst pain in the past 24 hours" Brief Pain Inventory (BPI) questions, scored daily in the patient's diary.

CONTACTS AND LOCATIONS:
Overall Officials: Alza Corporation Clinical Trial, Study Director — ALZA